CLINICAL TRIAL: NCT00998725
Title: A Pilot Study of Pharmacokinetic and Pharmacodynamic Activity of LoFemenal
Brief Title: Combined Oral Contraceptive (COC) Antiretroviral (ARV) Pharmacokinetics (PK) and Pharmacodynamics (PD) in Malawi
Acronym: COCARVPK
Status: Withdrawn | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Gretchen Stuart, MD, Associate Professor, University of North Carolina, Chapel Hill
Other Study IDs: 08-1500; AI050410 (#9p30) (Other: Merck)
Record Dates: First submitted 2009-10-16; First posted 2009-10-20 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Unintended Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- HIV+ARV+
- HIV+ARV-
- HIV negative

SUMMARY:
The purpose of this research study is to learn about the birth control pill called LoFemenal in HIV+ and HIV negative women who live in Malawi. This is a pilot study to determine the effect of antiretroviral therapy on the pharmacokinetics of the most commonly used oral contraceptive in HIV+ women; and to measure ovulation suppression in women taking the oral contraceptive pill and antiretroviral therapy at the same time. Nine women will be enrolled and will be followed for a total of 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Can provide informed consent
* Women ages 21-35 with known HIV status
* If HIV negative must have had an HIV test within the last 3 months
* Intend to stay in Lilongwe region for the duration of the study
* Desire to prevent pregnancy for at least the next six months
* Desires to use LoFemenal for contraception
* Has no known history of infertility
* Has intact uterus and at least one ovary
* Has regular monthly menses defined by menses occurring every 21-35 days
* Has not used another form of systemic hormonal contraception within the last six months.
* Has no contraindications to the combined oral contraceptive LoFemenal which include; any thrombophlebitis or thromboembolic disorders; cerebral-vascular or coronary-artery disease (current or history); thrombogenic valvulopathies; thrombogenic rhythm disorders; major surgery with prolonged immobilization; diabetes with vascular involvement; headaches with focal neurological symptoms; uncontrolled hypertension; known or suspected carcinoma of the breast or personal history of breast cancer; carcinoma of the endometrium or other known or suspected estrogen dependent neoplasia; undiagnosed abnormal genital bleeding; cholestatic jaundice of pregnancy or jaundice with prior pill use; hepatic adenomas or carcinomas or active lever disease, as long as liver function has not returned to normal; known or suspected pregnancy.

Exclusion Criteria:

* Hemoglobin < 10 mg/dL.
* Body mass index < 18.6 kg/m^2.
* Using any drugs known to interfere with cytochrome P450 system (such as rifampicin, phenytoin, carbamezapine, among others)
* In the opinion of the PI or study staff the individual cannot complete the study
* Cannot be adherent to other medications.

Additional inclusion criteria for the 3 HIV+ women on antiretroviral therapy:

* Must be on antiretroviral therapy which includes nevirapine for at least three consecutive months immediately prior to enrollment into the study
* Must report adherence to medication and medical visits
* Must be willing to use a barrier or backup method of contraception.

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 9 women with known HIV status who have regular monthly menses.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Number of women who complete the study | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen S Stuart, MD, MPHTM, Principal Investigator — University of North Carolina
Locations (1):
- UNC Project Malawi, Lilongwe, Malawi